CLINICAL TRIAL: NCT07073677
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Multi-center, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of IN-115314 Ointment in Mild to Moderate Atopic Dermatitis Adult Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of IN-115314 Ointment in Mild to Moderate Atopic Dermatitis Adult Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_JSI_201
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Mild to Moderate Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- J1 (Experimental): IN-115314 Ointment 1%
  Interventions: Drug: IN-115314 Ointment 1%
- J3 (Experimental): IN-115314 Ointment 3%
  Interventions: Drug: IN-115314 Ointment 3%
- PJ (Placebo Comparator): IN-115314 Ointment Placebo
  Interventions: Drug: IN-115314 Ointment placebo

INTERVENTIONS:
Drug: IN-115314 Ointment 1% — Twice daily(BID), for 56 day
  Arms: J1
Drug: IN-115314 Ointment 3% — Twice daily(BID), for 56 day
  Arms: J3
Drug: IN-115314 Ointment placebo — Twice daily(BID), IN-115314 Ointment Placebo for 28 days+ IN-115314 Ointment 3% for 28 days
  Arms: PJ

SUMMARY:
This study aims to evaluate the efficacy and safety of IN-115314 Ointment in mild to moderate atopic dermatitis adult patients

DETAILED DESCRIPTION:
1. Primary Objective

   - To evaluate the efficacy of IN-115314 ointment (1%, 3%) compared to placebo after multiple dosing, twice a day, in mild to moderate atopic dermatitis adult patients.
2. Secondary Objective

   * To evaluate the safety of IN-115314 ointment (1%, 3%) after multiple dosing, twice a day, in mild to moderate atopic dermatitis adult patients.
   * To evaluate the pharmacokinetic(PK) profile of IN-115314 ointment (1%, 3%) after multiple dosing ,twice a day, in mild to moderate atopic dermatitis adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers aged 19 or older when the informed consent is obtained.
2. Confirmed diagnosis of AD according the criteria of Hanifin and Rajka (1980).
3. AD lesions that can be applied by investigational product
4. AD diagnosed by EASI score of mild (EASI < 16) or moderate (16 ≤ EASI <

23) at screening. 5) Subjects who Investigator Global Assessment (IGA) of 2 to 3 at screening 6) Subjects who have a history of AD at least 12 months prior to screening and who have not improved or worsened the disease for at least one month prior to screening 7) Subjects who voluntarily decide to participate and agree to comply with the requirements

Exclusion Criteria:

1. Subjects who have the following prior/current history in addition to evidence or history of clinically significant skin disorders other than AD ( e.g., psoriasis, contact dermatitis, erythroderma)
2. Subjects who have the following prior/current history in addition to evidence or history of clinically significant skin disorders (e.g., hepatic, renal, Cardiovascular, respiratory, endocrine, neurological, hematological, immunological or immunodeficiency disease)
3. Subjects who have a history of malignant tumors within 5 years at screening (but, those who have passed five years without recurrence after active tumor treatment (surgery, chemotherapy, radiation therapy, etc.) can participate.)
4. Subjects who have clinically significant systemic or local skin infections or clinical signs of such infections within one week prior to the expeced initial application date (e.g., herpes simplex, shingles, chickenpox)
5. Subjects who have taken systemic anti-inflammatory for chronic or acute inflammatory disease within 2 weeks prior to the expected initial application date
6. Subjects who have a history of clinical significant hypersensitivity reactions to Investigational product , other drugs (aspirin, penicillin antibiotics, macrolide antibiotics, etc.) and moisturizers provided by sponsor (anaphylaxis or angioedema, etc.)
7. Subjects who have administered the following drugs within the specified period before the expected initial application date; subjects who are expected to be administered within the clinical trial period; subjects who are unable to stop administration Biological agents that may affect signs and symptoms of AD within 12 weeks (e.g., dupilumab)

   The following medications and treatments that may affect the signs and symptoms of atopic dermatitis within 4 weeks:
   * Systemic immunosuppressants/immunosuppressants
   * Oral Janus kinase (JAK) inhibitor medication
   * a live vaccine
   * systemic retinoid
   * phototherapy treatment
   * Systemic corticosteroids

   The following medications and treatments that may affect the signs and symptoms of atopic dermatitis within two weeks:
   * a systemic anti-inflammatory drug
   * systemic anti-microbial agents
   * bleach treatment

   The following medications that may affect the signs and symptoms of atopic dermatitis within one week:
   * topical corticosteroids
   * topical calcineurin inhibitor
   * topical antihistamines
   * a topical anti-microbial agent
   * a topical PDE-4 inhibitor
   * topical retinoid
   * Oral antihistamines
8. Subjects who have clinically significant findings on 12-lead ECG at screening
9. The following clinically significant findings on laboratory examination at screening

   * Hb < 10 g/dL
   * Platelet or ANC level < 0.5 x lower limit of normal
   * AST, ALT, ALP, γ-GTP is ≥ 2 or total bilirubin level is ≥ 1.5 x upper limit of normal;
   * Serum creatinine level is ≥ 2 x upper limit of normal;
   * Positive anti-HCV, HBs Ag, HIV Ag/Ab, or IGRA test.
10. Subjects who have uncontrolled hypertension (sitSBP ≥ 160 mmHg or sitDBP ≥ 100 mmHg)
11. Subjects who have history of drug or alcohol abuse in 56 weeks at screening
12. Subjects who have donated whole blood or apheresis within 4 weeks prior to the expected initial application date or received blood transfusion within 4 weeks prior to the expected initial application date, or subjects who cannot continuously abstain from blood donation over a period from the informed consent to PSV.
13. Subjects who have participated in other clinical trials within 4 weeks prior to the expected initial application date
14. Subjects who have scheduled surgery requiring hospitalization or requires surgical treatment over the clinical trial
15. Subjects or spouses (or partners) who have a plan for pregnancy or although unplanned pregnancy, are unable to use a highly effective method of contraception over a period from the informed consent to 90 days after the last dose of investigational product.
16. Pregnant or lactating woman
17. Naive in atopic dermatitis treatment
18. Subjects who are judged ineligible for the clinical study by the investigator due to reasons other than the above inclusion/exclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change rate in EASI score from the baseline after treatment | 4 weeks

SECONDARY OUTCOMES:
Change rate in EASI score from the baseline after treatment | 1 week, 2 weeks
Changes in EASI score from the baseline after treatment | 1 week, 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Son Sang Wook, Principal Investigator — Korea University Ansan Hospital

IPD SHARING:
Plan to Share IPD: No